CLINICAL TRIAL: NCT04068857
Title: Effects of Precuneus Repetitive Transcranial Magnetic Stimulation (rTMS) on Self-Referential Processing and Default Mode Network Functional Connectivity in Early Phase Psychosis
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) Self-Referential Processing (rTMS-SRP)
Acronym: rTMS-SRP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not going forward at this time.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Michael Francis, Associate Professor of Clinical Psychiatry, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1904511224
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia; Schizo Affective Disorder
Keywords: schizophrenia; schizoaffective disorder; psychosis; early phase
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- rTMS (Experimental)
  Interventions: Device: rTMS
- Sham (Sham Comparator)
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technique that received FDA clearance for use in treatment resistant major depressive disorder in 2008 and has become commonly used in clinical practice. rTMS utilizes the application of a repetitively pulsed magnetic field over the scalp to induce an electric field within a discrete area of the cerebral cortex. This electric field results in altered ion flow across the neuronal cellular membrane and ultimately changes in neuronal polarization. rTMS enables investigators to manipulate brain activity in a targeted cortical region as well as downstream connectivity within an associated neuronal circuit. High frequency (HF) rTMS leads to facilitatory effects on brain excitability. Previous studies have demonstrated that administration of as little as a single train or a small number of trains are able to produce an immediate increase in cortical excitability.

SUMMARY:
This will be a single site pilot study. 16 subjects with early phase psychosis (EPP), defined as medical record documentation of the onset of clinically significant psychotic symptoms within the past ten years, will be randomized 1:1 to double-blind treatment with 5 sessions of rTMS or sham stimulation directed at the bilateral precuneus over the course of 1 week. Subjects will undergo functional magnetic resonance imaging (fMRI) procedures, behavioral and cognitive assessments, and self-referential memory paradigm (SRMP) at baseline and immediately following the final rTMS or sham session. Contact with subjects will be conducted at two weeks after the end of study intervention for adverse event assessments. In the event new adverse events felt to be related to the study intervention have occurred following the termination of study procedures, subjects will be brought in for further safety assessments.

DETAILED DESCRIPTION:
A number of studies have investigated the therapeutic potential of rTMS in schizophrenia, noting improvements in treatment refractory auditory hallucinations as well as negative symptoms and cognitive dysfunction. However, no previous studies have examined the effects of precuneus directed rTMS on SRP deficits in schizophrenia. It is also important to note that the vast majority of studies using rTMS in schizophrenia have examined chronic populations where confounds associated with prolonged duration of illness may be present. Early phase psychosis (EPP) is a desirable population to study because these patients tend to have fewer psychiatric and physical comorbidities and less antipsychotic drug exposure, all of which are factors that may confound investigations of new treatment interventions for this illness. In light of the significant unmet medical need associated with schizophrenia and the grave clinical effect of disrupted SRP in the illness, rTMS modulating precuneus, and potentially DMN circuitry, represents an unexplored and potentially novel potential treatment option.

This study proposes to examine the application of rTMS targeting the precuneus for the treatment of disrupted SRP in EPP. This is an important population for study because if effective, rTMS may represent a preventative treatment for the development of poor outcomes and functioning associated with SRP deficits in in schizophrenia. This study will also seek to refine the understanding of the brain circuitry that mediates the potential pro-SRP effects of rTMS through the use of fMRI at baseline and following the course of rTMS administration.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 45 years of age
2. Within 10 years of illness onset as defined by entry into treatment for psychotic symptoms
3. Able to give informed consent
4. Willing and able to adhere to the study schedule
5. Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (SCID-5) diagnosis of schizophrenia or schizoaffective disorder
6. Clinical stability as defined by:

   * Clinical Global Impression scale - Severity (CGI-S) score of less than or equal to 4 (moderately ill) at baseline AND
   * No exacerbation of their illness within 4 weeks prior to randomization, leading to an intensification of psychiatric care in the opinion of the investigator. Examples of intensification of care include, but are not limited to: inpatient hospitalization, day/partial hospitalization, outpatient crisis management, or psychiatric treatment in an emergency room AND
   * Antipsychotic treatment stability for at least 4 weeks prior to randomization (no change in antipsychotic dosing or addition of any new antipsychotic medication).

Exclusion Criteria:

1. Lifetime history of a seizure, excluding febrile seizures and those induced by substance withdrawal
2. First degree relative (that is, biological father, mother, brother, sister, or child) with idiopathic epilepsy or other seizure disorder
3. History of significant neurological illness (including stroke, central nervous system (CNS) infection with persistent neurologic deficit, or other event deemed significant by PI)
4. History of head trauma as defined by a loss of consciousness or a post-concussive syndrome
5. Pregnant or breast feeding
6. Known intelligence quotient (IQ) < 70 based on subject report
7. Subjects with current acute, serious, or unstable medical conditions, including, but not limited to: inadequately controlled diabetes, asthma, chronic obstructive pulmonary disease (COPD), severe hypertriglyceridemia, recent cerebrovascular accidents, acute systemic infection or immunologic disease, unstable cardiovascular disorders, malnutrition, or hepatic, renal gastroenterological, respiratory, endocrine, neurologic, hematologic, or infectious diseases based on medical history or physical examination
8. Metallic objects planted in or near the head, including implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, transcutaneous electrical nerve stimulation (TENS) unit, ventriculoperitoneal shunt, or cochlear implants
9. Contraindications to MRI or otherwise unable to tolerate MRI procedures
10. History of electroconvulsive therapy
11. Subjects taking clozapine
12. Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to randomization
13. Subjects considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 90 days prior to screening
14. Current SCID-5 diagnosis of substance use disorder (excluding nicotine or caffeine)
15. Subjects who require concomitant treatment with prohibited medication, as specified in Attachment 2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
SRMP | 1 week
  To determine the effects of HF rTMS targeting the bilateral precuneus on SRP as measured by a self-referential memory paradigm (SRMP)
Default mode network functional connectivity (DMN FC) | 1 week
  To assess the effects of HF rTMS targeting the bilateral precuneus on DMN FC at rest

SECONDARY OUTCOMES:
Correlation between SRMP and DMN FC | 1 week
  Assessing the correlation between SRMP performance and DMN FC
SRMP and Scale to Assess Unawareness of Mental Disorder (SUM-D) | 1 week
  Assessing the correlation between SRMP performance and the SUM-D scale
SRMP and Beck Cognitive Insight Scale (BCIS) | 1 week
  Assessing the correlation between SRMP performance and the BCIS scale
SRMP and Birchwood Insight Scale | 1 week
  Assessing the correlation between SRMP performance and the Birchwood Insight Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Francis, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Center for Neuroimaging, Indianapolis, Indiana
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No